CLINICAL TRIAL: NCT06812507
Title: Evaluation of Placental Transfusion Techniques in of Prematurity Related Complications and Hematological Profile
Brief Title: Evaluation of Placental Transfusion Techniques in Prevention of Prematurity Related Complications and Effect on Their Hematological Profile
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Assistant professor of Pediatrics, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0107951
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Premature; Placental Transfusion
MeSH Terms: conditions — Premature Birth; Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The procedure of intact umbilical cord milking (I-UCM) (Experimental): Umbilical cord milking will be performed by holding the newborn at or
  ∼20 cm below the level of the placenta. The cord will be pinched between 2 fingers as close to the placenta as possible and milked toward the infant over a 2-second duration. The cord will then be released and allowed to refill with blood for a brief 1- to 2-second pause between each milking motion. This will be repeated for 2-4 times. After completion, the cord will be clamped, and the neonate will be handed to the resuscitation team.
  Interventions: Procedure: intact umbilical milking
- The procedure of Cut-umbilical cord milking(C-UCM): (Experimental): Another technique, used more often in Asia, involves clamping and cutting a long segment of the umbilical cord immediately at birth and passing the baby and the long cord to the pediatric provider, called C-UCM untwists the cord and milks the entire contents into the baby. Milking the cord 2-3 times before clamping may produce a similar placental transfusion as C-UCM
  Interventions: Procedure: cut umbilical milking
- The procedure of Delayed Cord Clamping (DCC): (Experimental): Infants placed on the maternal abdomen or at the introitus below the level of placenta and waiting at least 30- to 60-second before clamping the cord.
  Interventions: Procedure: Delayed cord clamping
- Control group: (No Intervention): patients will not receive any of the methods of placental transfusions

INTERVENTIONS:
Procedure: intact umbilical milking — Umbilical cord milking will be performed by holding the newborn at or
  ∼20 cm below the level of the placenta. The cord will be pinched between 2 fingers as close to the placenta as possible and milked toward the infant over a 2-second duration. The cord will then be released and allowed to refill with blood for a brief 1- to 2-second pause between each milking motion. This will be repeated for 2-4 times. After completion, the cord will be clamped, and the neonate will be handed to the resuscitation team.
  Arms: The procedure of intact umbilical cord milking (I-UCM)
Procedure: cut umbilical milking — Another technique, used more often in Asia, involves clamping and cutting a long segment of the umbilical cord immediately at birth and passing the baby and the long cord to the pediatric provider, called C-UCM untwists the cord and milks the entire contents into the baby. Milking the cord 2-3 times before clamping may produce a similar placental transfusion as C-UCM
  Arms: The procedure of Cut-umbilical cord milking(C-UCM):
Procedure: Delayed cord clamping — Infants placed on the maternal abdomen or at the introitus below the level of placenta and waiting at least 30- to 60-second before clamping the cord.
  Arms: The procedure of Delayed Cord Clamping (DCC):

SUMMARY:
The objective of this study is to evaluate the general course and prognosis associated with different methods of placental transfusion (Intact umbilical cord milking, cut- umbilical cord milking and delayed cord clamping) in premature neonates over the first days of life

ELIGIBILITY:
* Inclusion Criteria:

  1. Premature neonates ≤ 32 weeks gestational age regardless birth weight
  2. patients should be admitted to neonatal intensive care unit in the first day of life of life

Exclusion criteria:

* Exclusion Criteria:

Patient with any of the following will be excluded:

1. Major congenital anomalies (complex cyanotic heart disease, major central nervous system anomalies).
2. Evidence of head trauma causing major intracranial hemorrhage.
3. placental abnormalities like : abruptions, placenta previa or retroplacental hematoma.
4. Cord accident, or avulsion at the time of delivery.
5. Refusal to perform the intervention by the obstetrician

Ages: 1 Minute to 2 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | on admission (In first day after birth),as well as, at end of first , second and third weeks of lives
  hemoglobin level will be measured in gram/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Mohamed Farag, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request
Supporting Information: Study Protocol